CLINICAL TRIAL: NCT05884372
Title: Efficacy and Safety of Combination Denosumab With Eldecalcitol for Postmenopausal Women With Osteoporosis.(ESCORT)
Acronym: ESCORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xi'an Honghui Hospital (Other)
Collaborators: Chugai Pharma China Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Yuhong Zeng, Chief Physician, Xi'an Honghui Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELD-IIS00X
Record Dates: First submitted 2023-05-07; First posted 2023-06-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoporosis in Postmenopausal Women
MeSH Terms: interventions — eldecalcitol; Denosumab; Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab+Eldecalcitol (Experimental): Denosumab (subcutaneous injection 60mg/6 months) combined with ELD (oral 0.75μg/day) for 12 months.
  Interventions: Drug: Eldecalcitol; Drug: Denosumab
- Denosumab+Native Vitamin D+Calcium (Active Comparator): Denosumab (subcutaneous injection 60mg/6 months) combined with native vitamin D (oral 800IU/day) and Calcium (oral 600mg/day) for 12 months.
  Interventions: Drug: Native Vitamin D; Drug: Denosumab; Drug: Calcium

INTERVENTIONS:
Drug: Eldecalcitol — the same as arm descriptions.
  Arms: Denosumab+Eldecalcitol
Drug: Native Vitamin D — the same as arm descriptions.
  Arms: Denosumab+Native Vitamin D+Calcium
Drug: Denosumab — the same as arm descriptions.
Drug: Calcium — the same as arm descriptions.
  Arms: Denosumab+Native Vitamin D+Calcium

SUMMARY:
Primary objective:

To compare the bone mineral density (BMD) change under the treatment of denosumab with eldecalcitol or native vitamin D in postmenopausal women with osteoporosis on bone mineral density.

Secondary objective:

To compare the efficacy of denosumab with eldecalcitol or native vitamin D treatment in postmenopausal women with osteoporosis on bone turnover markers, serum PTH, serum calcium, serum phosphorus, muscle mass, muscle strength, body balance ability, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 1.Postmenopausal patients with osteoporosis, measured by dual energy X-ray absorptiometry (DXA), the T value of lumbar spine, femoral neck or total hip BMD is ≤-2.5, or with low mineral density (-2.5 < T-score < -1.0) plus a fragility fracture of the proximal humerus or distal forearm, or a history of vertebral compression fracture.
* 2.Voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

* 1.Suffering from hyperthyroidism, Cushing's syndrome, hypogonadism, poorly controlled diabetes mellitus (glycated hemoglobin [HbA1c>9.0%]), or other diseases that may lead to secondary osteoporosis.
* 2.Patients who have received denosumab therapy before screening: received oral bisphosphonate treatment more than 3 years or received bisphosphonate treatment within 6 months before screening, or received treatment with glucocorticoids, vitamin K, active vitamin D compounds, selective estrogen receptor modulators, calcitonin, hormone replacement therapy, or teriparatide within the 8 weeks prior to study enrollment..
* 3.Patients who at screening have urinary tract stones detected on B-mode ultrasonography or who have a prior history of urolithiasis.
* 4.Corrected serum calcium value at screening exceeds 2.6mmol/L (10.4mg/dL) or serum calcium value is lower than 2.12mmol/L(8 mg/dL) or hypercalciuria (> 0.4 mg/dL GF), or chronic kidney disease (eGFR < 30 mL/min/1.73 m2).
* 5.Patients with a history of malignant tumors.
* 6.Patients judged by investigators to be unsuitable as subjects.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
the percent change from baseline at month 12 in BMD at the lumbar spine L1-4. | 12 months
  the percent change from baseline at month 12 in BMD at the lumbar spine L1-4.

SECONDARY OUTCOMES:
the percent change from baseline at month 6 in BMD at the lumbar spine L1-4. | 6 months
  the percent change from baseline at month 6 in BMD at the lumbar spine L1-4.
the percent change from baseline at each visit in BMD at the femoral neck and total hip. | 12 months
  the percent change from baseline at each visit in BMD at the femoral neck and total hip.
the percent change from baseline at each visit in serum CTX,P1NP,PTH. | 12 months
  the percent change from baseline at each visit in serum CTX,P1NP,PTH.
the score change from baseline at month 6 and month 12 in quality of life by 16-item Assessment of Health-Related Quality of Life in Osteoporosis,(ECOS-16). | 12 months
  the score change from baseline at month 6 and month 12 in quality of life by 16-item Assessment of Health-Related Quality of Life in Osteoporosis,(ECOS-16). The scale ranges from 16 to 80, with higher scores meaning higher risk.
Incidence rate of new vertebral fracture and new non-vertebral fracture in 1 year. | 12 months
  Incidence rate of new vertebral fracture and new non-vertebral fracture in 1 year.

OTHER OUTCOMES:
the change from baseline at month 6 and month 12 in body balance ability by measuring One Leg Standing (OLS). | 12 months
  the change from baseline at month 6 and month 12 in body balance ability by measuring One Leg Standing (OLS).
the change from baseline at month 6 and month 12 in limb skeletal muscle content by DXA. | 12 months
  the change from baseline at month 6 and month 12 in limb skeletal muscle content by DXA.
the change from baseline at month 6 and month 12 in physical function by measuring 5 times chair stand. | 12 months
  the change from baseline at month 6 and month 12 in physical function by measuring 5 times chair stand.
the change from baseline at month 6 and month 12 in muscle strength by measuring handgrip strength. | 12 months
  the change from baseline at month 6 and month 12 in muscle strength by measuring grip strength.
the change from baseline at month 6 and month 12 in body balance ability by measuring 10 Meter Walk (10MW). | 12 months
  the change from baseline at month 6 and month 12 in body balance ability by measuring 10 Meter Walk (10MW).
the change from baseline at month 6 and month 12 in body balance ability by measuring Timed Up and Go (TUG). | 12 months
  the change from baseline at month 6 and month 12 in body balance ability by measuring Timed Up and Go (TUG).

CONTACTS AND LOCATIONS:
Locations (1):
- Zeng,Yuhong, Xi'an, China

IPD SHARING:
Plan to Share IPD: No